CLINICAL TRIAL: NCT05795439
Title: The CARING Study: Creating and Restoring Health Through Nutrition Guidance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Collaborators: Blue Cross Blue Shield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00069695
Record Dates: First submitted 2023-03-08; First posted 2023-04-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Type2diabetes; Type 2 Diabetes Treated With Insulin
Keywords: Diabetes; Type2; Insulin; A1C
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Diet, Fat-Restricted; Diet, Vegan

STUDY DESIGN:
Intervention Model Description: One arm, the intervention group, will be randomly assigned to be on a low-fat vegan diet for the duration of the study. The other arm, the control group, will maintain their pre-study diet for the duration of the study.
Who Masked: Investigator
Masking Description: The control group will be asked to stay on their usual diet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The Intervention group arm of participants will be asked to attend weekly online classes on nutrition and health and to follow a low-fat, vegan diet for 16 weeks.
  Interventions: Behavioral: Low-fat, vegan diet
- Control Group (No Intervention): The Control group arm of participants will be asked to maintain their regular, pre-study diet.

INTERVENTIONS:
Behavioral: Low-fat, vegan diet — The intervention diet consists of whole grains, vegetables, legumes, and fruits, with no restriction on energy intake. Participants will also be guided to favor foods with a low glycemic index. Animal products and added oils will be excluded. The diet is designed to derive approximately 10% of energy from fat, approximately 10-15% of energy from protein, and the remainder from mostly complex carbohydrates. The diet will also provide approximately 40 g of fiber per day.
  Arms: Intervention Group

SUMMARY:
The CARING study assesses the health benefits of nutrition education for Blue Cross Blue Shield subscribers, as well as potential healthcare cost savings to subscribers and the insurance company.

DETAILED DESCRIPTION:
Among Blue Cross Blue Shield subscribers, individuals with type 2 diabetes will be randomly selected and invited to participate in an interventional trial. A control group matched for relevant variables will be selected from Blue Cross Blue Shield subscribers.

The Intervention group participants will be asked to attend weekly online classes on nutrition and health and to follow a low-fat, vegan diet for 16 weeks. Body weight, plasma lipids, HbA1C, dietary intake and adherence, and food acceptability will be assessed at baseline and at 16 weeks. Their longer-term medical utilization will then be tracked for another 2 years and compared with that of a control population selected from Blue Cross Blue Shield subscribers. Weekly classes will be offered for the whole 2-year follow-up period. Plasma lipids and HbA1C will be assessed every 6 months during the 2-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Blue Cross Blue Shield subscriber continuously enrolled for the prior 12 months
2. Male or female
3. Age at least 18 years
4. Have a diagnosis of type 2 diabetes
5. Ability and willingness to participate in all components of the study, including:

   1. Following a plant-based diet for the initial 16 weeks of the study;
   2. Attending weekly online classes for the initial 16 weeks of the study; and
   3. Keeping physical activity level consistent throughout the initial 16 weeks of the study.

Exclusion Criteria:

1. Diabetes mellitus type 1 or history of any endocrine condition that would affect body weight, such as a pituitary abnormality or Cushing's syndrome
2. Smoking during the past six months
3. Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
4. Current or unresolved past drug abuse
5. Recently gave birth, pregnant, or plans to become pregnant before or during the study period
6. Unstable medical or psychiatric status
7. Cancer diagnosis
8. Chronic kidney disease, stage 4 or 5
9. Evidence of an eating disorder
10. Lack of English fluency
11. Bariatric surgery in the last 6 months
12. Dementia
13. Institutional custodial care
14. End of life
15. Palliative Care
16. Actively engaged in specific BCBSM diabetes programs and case management programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Medical Utilization | 16 weeks, 1 year, and 2 years
  This study will assess the effectiveness of a series of plant-based nutrition classes on health changes, measured by combined subscriber and insurance total cost of care (healthcare and health benefits).
Body Weight | 16 weeks, 1 year, and 2 years
  This study will assess the association of attending a series of plant-based nutrition classes with pre-post changes in body weight.
Plasma Lipid Concentrations | 16 weeks, Every 6 months during the 2-year follow-up period
  This study will assess the association of attending a series of plant-based nutrition classes with pre-post changes in plasma lipid concentrations.
HbA1C | 16 weeks, Every 6 months during the 2-year follow-up period
  This study will assess the association of attending a series of plant-based nutrition classes on with pre-post changes in glycemic control in individuals with type 2 diabetes as assessed by hemoglobic A1c (HbA1c) and use of medications.

SECONDARY OUTCOMES:
Diet Acceptability | 16 weeks
  In addition, this study will assess the impact of association of attending a series of plant-based nutrition classes on pre-post changes in diet acceptability. Diet acceptability will be determined using the Food Acceptability Questionnaire (FAQ), asking participants to think about foods they have consumed in the prior two weeks to taking the FAQ, where higher scores indicate greater acceptability. There are eleven questions ranking answers on a scale of 1-7, and one question ranking answers on a scale from 1-13.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Barnard, MD, Principal Investigator — Physicians Committee for Responsible Medicine
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hales CM, Carroll MD, Fryar CD, Ogden CL. Prevalence of Obesity and Severe Obesity Among Adults: United States, 2017-2018. NCHS Data Brief. 2020 Feb;(360):1-8. PMID 32487284
- [Background] Pi-Sunyer X. The medical risks of obesity. Postgrad Med. 2009 Nov;121(6):21-33. doi: 10.3810/pgm.2009.11.2074. PMID 19940414
- [Background] Viguiliouk E, Kendall CW, Kahleova H, Rahelic D, Salas-Salvado J, Choo VL, Mejia SB, Stewart SE, Leiter LA, Jenkins DJ, Sievenpiper JL. Effect of vegetarian dietary patterns on cardiometabolic risk factors in diabetes: A systematic review and meta-analysis of randomized controlled trials. Clin Nutr. 2019 Jun;38(3):1133-1145. doi: 10.1016/j.clnu.2018.05.032. Epub 2018 Jun 13. PMID 29960809
- [Background] Esselstyn CB Jr. Updating a 12-year experience with arrest and reversal therapy for coronary heart disease (an overdue requiem for palliative cardiology). Am J Cardiol. 1999 Aug 1;84(3):339-41, A8. doi: 10.1016/s0002-9149(99)00290-8. PMID 10496449
- [Background] Esselstyn CB Jr, Ellis SG, Medendorp SV, Crowe TD. A strategy to arrest and reverse coronary artery disease: a 5-year longitudinal study of a single physician's practice. J Fam Pract. 1995 Dec;41(6):560-8. PMID 7500065
- [Background] Ornish D, Brown SE, Scherwitz LW, Billings JH, Armstrong WT, Ports TA, McLanahan SM, Kirkeeide RL, Brand RJ, Gould KL. Can lifestyle changes reverse coronary heart disease? The Lifestyle Heart Trial. Lancet. 1990 Jul 21;336(8708):129-33. doi: 10.1016/0140-6736(90)91656-u. PMID 1973470
- [Background] Tonstad S, Butler T, Yan R, Fraser GE. Type of vegetarian diet, body weight, and prevalence of type 2 diabetes. Diabetes Care. 2009 May;32(5):791-6. doi: 10.2337/dc08-1886. Epub 2009 Apr 7. PMID 19351712
- [Background] Schepers J, Annemans L. The potential health and economic effects of plant-based food patterns in Belgium and the United Kingdom. Nutrition. 2018 Apr;48:24-32. doi: 10.1016/j.nut.2017.11.028. Epub 2017 Dec 15. PMID 29469016
- [Background] Craig WJ, Mangels AR; American Dietetic Association. Position of the American Dietetic Association: vegetarian diets. J Am Diet Assoc. 2009 Jul;109(7):1266-82. doi: 10.1016/j.jada.2009.05.027. PMID 19562864
- [Background] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Background] Hernan MA, Robins JM. Per-Protocol Analyses of Pragmatic Trials. N Engl J Med. 2017 Oct 5;377(14):1391-1398. doi: 10.1056/NEJMsm1605385. No abstract available. PMID 28976864